CLINICAL TRIAL: NCT06844071
Title: The Sentio System: Post-market Evaluation of Safety and Performance in Adolescents With Mixed/Conductive Hearing Loss and Single Sided Deafness
Brief Title: The Sentio System: Post-market Evaluation of Safety and Performance in Adolescents
Status: Recruiting | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BC120
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- subjects

SUMMARY:
This study is a post-market, multicentre, prospective, single arm investigation aimed to systematically collect safety and performance data on the Sentio system, when used as intended for adolescents (12-17 years inclusive).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria to be eligible for participation in the investigation:

  1. Signed Informed Consent Form (signed by parent or legal guardian and child).
  2. Subjects aged 12 to 17 years of age (inclusive)
  3. Subjects with the following audiometric criteria consistent with the current and approved labeling of the device:

     3.1 Conductive or mixed hearing loss with a pure tone average (PTA) bone conduction (BC) threshold (measured at 0.5, 1, 2, and 3 kHz) of the indicated ear better than or equal to 45 dB HL.

     3.2 OR subjects with a profound sensorineural hearing loss in one ear and normal hearing in the opposite ear (i.e., single-sided deafness or "SSD"). The pure tone average air conduction hearing (AC) thresholds of the hearing ear should be better than or equal to 20 dB HL (measured at 0.5, 1, 2, and 3 kHz).

     3.3 OR subjects who are indicated for an air-conduction contralateral routing of signals (AC CROS) hearing aid, but who for some reason cannot or will not use an AC CROS.
  4. Prior experience with amplified sound through properly fitted amplification devices such as a hearing aid, a CROS device, or a non-surgical bone conduction solution (e.g., a softband or sound arc).
  5. For patients with conductive or mixed hearing losses sufficient (e.g., >25 dB) air bone gap (ABG) at the ear to be implanted.
  6. Subjects and parent(s) or legal guardian have the ability and willingness to comply with all investigational procedures/requirements, as determined by the Investigator.

Exclusion Criteria:

* Subjects meeting any of the following criteria will not be permitted to participate in the investigation:

  1. Medical condition(s) that contraindicates implant surgery or anesthesia.
  2. Untreated ongoing middle ear infection at the time of surgery.
  3. Known or suspected contact allergy to silicone or other material used in the Sentio system.
  4. Insufficient bone quality/quantity/depth or skull size for implantation of a Sentio Ti implant, assessed according to clinical practice.
  5. Known conditions that could jeopardize wound healing and skin condition e.g. uncontrolled diabetes over time or skin or scalp condition(s) that may preclude attachment to, or interfere with usage of, the sound processor as judged by the investigator.
  6. Subject that has received radiotherapy in the area of implantation or is planned for such radiotherapy or similar during the investigation period.
  7. For bilateral asymmetric* candidates, subjects already treated with a bone-anchored hearing solution on the side with the best BC thresholds.
  8. Known chronic or non-revisable vestibular or balance disorder.
  9. Known abnormally progressive sensorineural hearing loss.
  10. Currently participating, or participated within the last 30 days, in another clinical investigation involving an investigational drug or device that could impact the safety or effectiveness of the Sentio system as determined by the investigator.
  11. Use of active implantable or body worn devices that for medical reasons cannot be removed or discontinued, such as CSF shunts, implantable cardiac pacemakers, defibrillators, or neurostimulators.
  12. Known need for frequent MRI investigations for follow-up of other diseases.
  13. Current or known future use of ototoxic drugs that could be harmful to the hearing, as judged by the investigator.
  14. Known retro cochlear pathology and auditory processing disorders that may have an impact on the outcome of the investigation.
  15. Any other known condition (e.g., developmental or learning delay or disability) that the investigator determines could interfere with compliance or investigation assessments.
  16. Any subject that according to the Declaration of Helsinki is deemed unsuitable for enrollment.

      * Defined as >10 dB difference measured across PTA of .5, 1, 2, & 3kHz

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The investigation population will be comprised of the main patient groups indicated for the Sentio system: patients with either conductive/mixed hearing loss, SSD patients, or patients who for some reason cannot or will not use an AC CROS. The Sentio system is indicated for patients above the age of 12 and the investigation population will enroll adolescents between 12-17 years.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
A. To demonstrate that the Sentio system improves hearing on the implanted ear. | 3months post implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Atlanta Institute for ENT, Atlanta, Georgia, United States